CLINICAL TRIAL: NCT05694494
Title: Training- and Cost-effectiveness of an Internet-based Lifestyle-integrated Functional Exercise Program (iLiFE) on Reducing Falls, and Promoting Exercise Adherence in Community Older Fallers: a Randomized Controlled Trial
Brief Title: Training- and Cost-effectiveness of an Internet-based Lifestyle-integrated Functional Exercise Program (iLiFE)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Timothy Kwok, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020.622-T
Record Dates: First submitted 2023-01-03; First posted 2023-01-23 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Fall

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iLiFE (Experimental): receiving Lifestyle-integrated Functional Exercise training and home safety assessment
  Interventions: Behavioral: internet-based Lifestyle-integrated Functional Exercise (iLiFE)
- attention control (Placebo Comparator): upper limb exercise training
  Interventions: Behavioral: upper limb exercise training

INTERVENTIONS:
Behavioral: internet-based Lifestyle-integrated Functional Exercise (iLiFE) — receiving internet-based LiFE training and home safety assessment
  Arms: iLiFE
Behavioral: upper limb exercise training — upper limb exercise training
  Arms: attention control

SUMMARY:
Falls are the second leading cause of unintentional injury and death around the globe. About one in every three older adults falls each year worldwide. With the aging population, the cost of treating fall-related injuries is increasing exponentially. There is a pressing need for a cost-effective fall prevention program. Ample evidence has shown the substantial standalone effectiveness of well-designed physical exercises in preventing falls. However, continuous exercise adherence is required for a long-lasting fall prevention effect. Unfortunately, adherence to an exercise program was generally only 21%. Building up the habit of doing regular exercise is thus crucial in preventing falls. Lifestyle integrated Functional Exercise program (LiFE) has been shown to be able to reduce the fall rate by 31% and maintain 64% of the participants exercising at 12 months follow-up. This proposed randomized controlled trial aims at comparing the effectiveness of an internet-based LiFE in reducing subsequent falls and promoting exercise adherence in community-dwelling older adults.

DETAILED DESCRIPTION:
All subjects will then be randomly assigned to receive either an internet-based therapist-led LiFE program with a home environment safety assessment (iLiFE) or attention control intervention. Randomization into block groups of four in a 1:1 ratio (the iLiFE group or the attention control group) will be generated in a password-protected excel file by independent research personnel not involved in data collection or intervention after the baseline assessment. The randomization will be concealed by the independent personnel. Research assistants who are blinded to the group allocation will conduct all the subsequent monthly surveillance and assessments at baseline and follow-up sessions. All data will also be entered and checked by the blinded research assistants. All procedures concur with the Declaration of Helsinki (2013).

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 65 years,
* community-dwelling,
* have a fall history in the previous 12 months,
* have a moderate or above risk of falls as assessed by the Physiological Profile Assessment (total z-score ≥ 1)
* can ambulate on level surfaces without physical contact of another person as assessed by Functional Ambulation Category (score ≥ 3)
* cognitively intact as assessed by the Hong Kong version of the Montreal Cognitive Assessment-5-minute protocol (score ≥ 16th percentile of the age and education-adjusted cut-off score)
* able to communicate effectively.

Exclusion Criteria:

* uncorrected vision or hearing impairment,
* unstable medical condition that may preclude the planned exercises, and
* have been receiving or planning to receive any fall prevention program within the study period.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 322 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
fall incidence as assessed by monthly telephone or internet follow-up | 12 months

SECONDARY OUTCOMES:
physiological fall risk as assessed by the Physiological Profile Assessment (PPA) | 4 months
  will be done at the baseline- and re-assessments
balance as assessed by the 4-stage stance | 4 months
  will be done at the baseline- and re-assessments
balance as assessed by functional reach tests | 4 months
  will be done at the baseline- and re-assessments
mobility as assessed by the Short Physical Performance Battery Test | 4 months
  will be done at the baseline- and re-assessments
mobility as assessed by the Timed Up and Go Test | 4 months
  will be done at the baseline- and re-assessments
mobility as assessed by the Ten Metre Walk Test | 4 months
  will be done at the baseline- and re-assessments
muscle mass as assessed by the Bioimpedance Analysis (BIA) | 4 months
  will be done at the baseline- and re-assessments
postural hypotension as assessed by the blood pressure in sitting and standing | 4 months
  will be done at the baseline- and re-assessments
physical activity level as assessed by thigh-worn accelerometer (ActivPAL4 physical activity monitor, PAL Technologies Ltd., Glasgow, UK) | 4 months
  The participants will be required to wear the device for 7 consecutive days right after the baseline assessment and the re-assessment. Data about the duration of time spent in different activity types such as walking and sitting will be extracted and calculated on a daily basis.
Cognitive flexibility as assessed by Trail Making Test | 4 months
  will be done at the baseline- and re-assessments
balance confidence as assessed by the Short version of the Chinese version of the Activities-specific Balance Confidence Scale | 12 months
  will be done at the baseline assessment, re-assessment, and the last monthly telephone or internet follow-up. The participants will be asked to indicate their level of confidence in performing each activity on a 0-100 scale. A higher score indicates better balance confidence.
exercise adherence as assessed by Section B of the Exercise Adherence Rating Scale | 12 months
  This will be done at the re-assessment and the last monthly telephone or internet follow-up. The total score ranges from 0 to 24. Higher total scores indicate better exercise adherence.
health-related quality of life as assessed by EQ-5D-5L | 12 months
  will be done at the baseline and re-assessment and the last monthly telephone or internet follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Kwok, Principal Investigator — The Chinese Univsersity of Hong Kong
Locations (1):
- The Chinese University of Hong Kong Jockey Club Centre for Osteoporosis Care and Control, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No